CLINICAL TRIAL: NCT02565784
Title: An Open, Evaluator-blinded, Non-comparative, Multi-center Study to Assess the Safety and Efficacy of Restylane Lidocaine and Restylane Perlane Lidocaine for Facial Augmentation in Asian Population
Brief Title: Safety and Efficacy of Restylane Lidocaine and Restylane Perlane Lidocaine for Facial Augmentation in Asian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05DF1315
Record Dates: First submitted 2015-09-23; First posted 2015-10-01 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intradermal injection (Experimental): Restylane and/or Perlane
  Interventions: Device: Restylane; Device: Perlane

INTERVENTIONS:
Device: Restylane — Facial tissue augmentation
Device: Perlane — Facial tissue augmentation

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Restylane Lidocaine and Restylane Perlane Lidocaine after the first and second treatment when used for facial augmentation in Asian population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects intent to undergo facial filler treatment for either volume loss or contouring
* Subjects requiring treatment in two to four of pre-defined areas in the face (upper cheeks, nasolabial folds, temples, nose and chin)
* Require 3-5 ml of investigational products to achieve a clinically meaningful improvement in appearance
* Facial appearance as Han Chinese
* Non-pregnant, non-breast feeding female
* Signed informed consent

Exclusion Criteria:

* Previous facial surgery (e.g. rhinoplasty) or permanent implant in the area to be treated.
* History of chronic sinusitis or rhinitis (only applicable for subjects injected in the nose).
* Subjects who needs to use heavy glasses during the study (only applicable for subjects injected in the nose).
* Previous tissue augmenting therapy or contouring with permanent filler or fat injection in the facial area.
* Previous treatment with Hyaluronic acid (HA) fillers or Restylane Skinboosters in the facial area within 12 months before treatment.
* Previous treatment with non-HA fillers such as CaHA (Calcium Hydroxylapatite) or PLLA (Poly L-Lactic Acid) within 24 months before treatment.
* Previous revitalization with neurotoxin in the facial area within six (6) months before treatment.
* Previous tissue revitalization treatment with laser or light, mesotherapy, chemical peeling or dermabrasion in the facial area within six (6) months before treatment.
* Any medical condition that, in the opinion of the investigator, would make the subject unsuitable for inclusion (e.g. a chronic, relapsing or hereditary disease that may interfere with the outcome of the study).

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12-29 (Actual); Study Completion 2018-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Q-Med AB, Study Director — Galderma R&D
Locations (2):
- Taiwan (2):
  - Galderma Research Site, Kaohsiung City
  - Galderma Research Site, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Treatment
Arm/Group | Intradermal Injection
Started | 100
6 Months Follow-up | 99
12 Months Follow-up | 98
Completed | 98
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: Second Treatment
Arm/Group | Intradermal Injection
Started | 98
6 Months Follow-up | 97
12 Months Follow-up | 96
Completed | 96
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intradermal Injection
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Improved in "Global Facial Aesthetic Appearance" - Judged by Participant
Description: Number of improved participants according to Global Aesthetic Improvement Scale (GAIS) 6 months after initial treatment.
  The GAIS is a qualitative 5-graded scale evaluating aesthetic improvement: Very much improved, Much improved, Improved, No change, Worse.
  A participant is considered "improved" if she answers Very much improved, Much improved, or Improved.
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intradermal Injection
Number analyzed (Participants) | 99
percentage of participants | 95 [89 to 98]

2. Secondary Outcome: Percentage of Participants Improved in Nasolabial Fold Severity (Merz Aesthetic Scale) - Judged by Investigator
Description: The Merz aesthetic scale for nasolabial folds (NLFs) is a validated photograph-based outcome instrument designed specifically for assessment of NLFs. The scale is graded 0-4 where 0 is "No folds" and 4 is "Very severe folds".
  A participant is considered improved if she scores at least one grade improvement from baseline.
Time Frame: 6 and 12 Months after first and second treatment, respectively
Population: In total, 88 participants were injected in the right NLF and 86 participants were injected in the left NLF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Right Nasolabial Fold; Left Nasolabial Fold: Intradermal injection
  Restylane and/or Perlane
  Restylane: Facial tissue augmentation
  Perlane: Facial tissue augmentation
Arm/Group | Right Nasolabial Fold | Left Nasolabial Fold
Number analyzed (Participants) | 88 | 86
percentage of participants
  6 Months after first treatment: number analyzed (Participants) | 87 | 86
  6 Months after first treatment | 54 [43 to 65] | 65 [54 to 75]
  12 Months after first treatment: number analyzed (Participants) | 86 | 85
  12 Months after first treatment | 47 [36 to 58] | 46 [35 to 57]
  6 Months after second treatment: number analyzed (Participants) | 85 | 84
  6 Months after second treatment | 65 [54 to 75] | 62 [51 to 72]
  12 Months after second treatment: number analyzed (Participants) | 84 | 83
  12 Months after second treatment | 54 [42 to 65] | 55 [44 to 66]

3. Secondary Outcome: Percentage of Participants Improved in Upper Cheek Fullness - Judged by Investigator
Description: The Merz aesthetic scale for upper cheek fullness is a validated photograph-based outcome instrument designed specifically for assessing cheek fullness. The scale is graded 0-4 where 0 is "Full upper cheek" and 4 is "Very severely sunken upper cheek".
  A participant is assessed as improved if she scores at least one grade improvement from baseline.
Time Frame: 6 and 12 Months after first and second treatment, respectively
Population: All 100 participants were injected in the upper cheeks, but 1 participant was not injected in left upper cheek at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Right Upper Cheek; Left Upper Cheek: Intradermal injection
  Restylane and/or Perlane
  Restylane: Facial tissue augmentation
  Perlane: Facial tissue augmentation
Arm/Group | Right Upper Cheek | Left Upper Cheek
Number analyzed (Participants) | 100 | 99
percentage of participants
  6 Months after first treatment: number analyzed (Participants) | 99 | 98
  6 Months after first treatment | 66 [55 to 75] | 67 [57 to 77]
  12 Months after first treatment: number analyzed (Participants) | 98 | 97
  12 Months after first treatment | 38 [28 to 48] | 43 [33 to 54]
  6 Months after second treatment: number analyzed (Participants) | 97 | 96
  6 Months after second treatment | 77 [68 to 85] | 78 [69 to 86]
  12 Months after second treatment: number analyzed (Participants) | 96 | 95
  12 Months after second treatment | 69 [59 to 78] | 71 [60 to 79]

ADVERSE EVENTS:
Time Frame: 2 years, 4 months
Description: Each subject was to be questioned about AEs at each study visit following the Screening Visit.
  The question to be asked was:"Since your last clinical visit have you had any health problems?" Information on AEs could also be obtained from signs and symptoms detected during an examination or from a laboratory test, observations made by the study site personnel, subject diaries, or spontaneous reports from subjects or their relatives.
Arm/Group | Intradermal Injection
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 5/100
Other Adverse Events (participants affected / at risk) | 34/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intradermal Injection (N=100)
Chronic paranasal sinusitis (Infections and infestations) | 1 (1)
Herpes simplex progenitalis (Infections and infestations) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intraductal papilloma (benign) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Left ovary tumor with endometrial polyps (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intradermal Injection (N=100)
Nasopharyngitis (Infections and infestations) | 18 (24)
Upper respiratory tract infection (Infections and infestations) | 10 (13)
Acne (Skin and subcutaneous tissue disorders) | 6 (10)
Implant site bruising (General disorders) | 6 (7)
Implant site pain (General disorders) | 5 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes